CLINICAL TRIAL: NCT05210946
Title: A Single-Arm Clinical Study of Pemigatinib in the Treatment of Advanced Non-Small Cell Lung Cancer Patients With FGFR Gene Alterations Who Have Failed Standard Therapy
Brief Title: A Single-Arm Clinical Study of Pemigatinib in the Treatment of Advanced Non-Small Cell Lung Cancer Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Principal Investigator, Huang Jianan, Chief physician， Director of the Department of Respiratory and Critical Care Medicine at the First Affiliated Hospital of Soochow University, The First Affiliated Hospital of Soochow University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIBI375Y005
Record Dates: First submitted 2022-01-14; First posted 2022-01-27 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pemigatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pemigatinib in Advanced Non-Small Cell Lung Cancer Patients with FGFR Gene Alterations (Experimental): This study is a prospective single-arm clinical study. Advanced non-small cell lung cancer patients with known FGFR 1-3 alterations (including but not limited to FGFR amplification, rearrangement/fusion, mutation, etc.) who have failed standard therapy will be enrolled in this study once they have signed the informed consent form (ICF) and been identified as eligible in screening. The patients will receive 13.5 mg of pemigatinib once a day (QD) orally following a 2-week administration/
  1-week interruption regimen. They will be dosed until disease progression or intolerable toxicity. During treatment, clinical tumor imaging evaluation will be performed according to RECIST v1.1 every 6 weeks (± 7 days) and then every 9 weeks (± 7 days) after week 48. Safety will be assessed according to
  Interventions: Drug: Pemigatinib

INTERVENTIONS:
Drug: Pemigatinib — Advanced non-small cell lung cancer patients with known FGFR 1-3 alterations (including but not limited to FGFR amplification, rearrangement/fusion, mutation, etc.) who have failed standard therapy will be enrolled in this study once they have signed the informed consent form (ICF) and been identified as eligible in screening. The patients will receive 13.5 mg of pemigatinib once a day (QD) orally following a 2-week administration/
  1-week interruption regimen. They will be dosed until disease progression or intolerable toxicity. During treatment, clinical tumor imaging evaluation will be performed according to RECIST v1.1 every 6 weeks (± 7 days) and then every 9 weeks (± 7 days) after week 48. Safety will be assessed according to NCI-CTCAE 5.0.

SUMMARY:
Primary objective:

● To evaluate the efficacy of pemigatinib in advanced non-small cell lung cancer patients with fibroblast growth factor receptor 1-3 (FGFR 1-3) alterations (including but not limited to FGFR amplification, rearrangement/fusion, mutation, etc.) who have failed standard therapy.

Secondary objective:

● To evaluate the safety and tolerability of pemigatinib in advanced non-small cell lung cancer patients with known FGFR 1-3 alterations (including but not limited to FGFR amplification, rearrangement/fusion, mutation, etc.) who have failed standard therapy, including the incidence of adverse events (AEs) and serious adverse events (SAEs), as well as the incidence of AEs/SAEs resulting in treatment discontinuation.

DETAILED DESCRIPTION:
This study is a prospective single-arm clinical study. Advanced non-small cell lung cancer patients with known FGFR 1-3 alterations (including but not limited to FGFR amplification, rearrangement/fusion, mutation, etc.) who have failed standard therapy will be enrolled in this study once they have signed the informed consent form (ICF) and been identified as eligible in screening. The patients will receive 13.5 mg of pemigatinib once a day (QD) orally following a 2-week administration/

1-week interruption regimen. They will be dosed until disease progression or intolerable toxicity. During treatment, clinical tumor imaging evaluation will be performed according to RECIST v1.1 every 6 weeks (± 7 days) and then every 9 weeks (± 7 days) after week 48. Safety will be assessed according to NCI-CTCAE 5.0.

ELIGIBILITY:
Inclusion Criteria:

Subjects must sign a written ICF prior to the implementation of any procedures related to the study;

1. Aged ≥ 18 years old;
2. Patients with histologically or cytologically confirmed unresectable stage IIIB-IIIC or stage IV NSCLC (staged according to the 8th Edition of the TNM Classification for Lung Cancer published by the International Association for the Study of Lung Cancer and American Joint Committee on Cancer);
3. Have at least one measurable lesion according to RECIST v1.1;
4. With histologically confirmed FGFR 1-3 alterations, including but not limited to amplification, mutation, fusion/rearrangement, etc.;
5. Have failed second-line and above standard therapies. Patients who have EGFR-sensitive mutations or are positive for ALK/ROS1 rearrangements shall receive at least one line of EGFR/ALK/ROS1 inhibitor treatment (Patients with EGFR-sensitive mutations who have received a first- or second-generation TKI should fail the treatment with a third-generation TKI (e.g., osimertinib) if they are positive for T790M mutations); Note: Patients who have a relapse within 6 months after a radical surgery or radical concurrent chemoradiotherapy can be enrolled if they have failed at least one line of systematic therapy after the relapse.
6. No previous use of small molecule multi-target drugs targeting the FGFR pathway (including anlotinib, lenvatinib, sorafenib, apatinib, bevacizumab, Endostar, etc.);
7. ECOG physical performance status score of 0-1;
8. Expected survival time > 3 months;
9. Patients with brain metastases who are asymptomatic or have stable symptoms after locoregional treatment can be enrolled as long as they:

1) Have measurable lesions outside the central nervous system; 2) Have no central nervous system symptoms or no aggravation of symptoms for at least 2 weeks; 3) Do not need glucocorticoid treatment or stop glucocorticoid treatment within 7 days before the first dose of the investigational drug.

10. Patients who have completed palliative radiotherapy one week prior to study enrollment with their radiotherapy-related toxicity reduced to grade 1 or lower (CTCAE5.0) can be enrolled.

11. For evidence of sufficient organ functions, the subjects shall meet the following laboratory parameters:

1. Absolute neutrophil count (ANC) ≥ 1.5 × 109/L without use of granulocyte colony stimulating factor in recent 14 days;
2. Platelet count ≥ 100 × 109/L without blood transfusion in recent 14 days;
3. Hemoglobin > 9 g/dL without blood transfusion or erythropoietin use in recent 14 days;
4. Total bilirubin ≤ 1.5 × upper limit of normal (ULN); or total bilirubin

   > ULN, direct bilirubin ≤ ULN;
5. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT)

   ≤ 2.5 × ULN (ALT or AST ≤ 5 × ULN for patients with liver metastasis);
6. Blood creatinine ≤ 1.5 × ULN and creatinine clearance (calculated by Cockcroft-Gault formula) ≥ 50 mL/min;
7. Good coagulation function: international normalized ratio (INR) or prothrombin time (PT) ≤ 1.5 × ULN. (For subjects receiving an anticoagulant therapy, PT within the range proposed for the anticoagulant drug is acceptable).

12. Women of childbearing potential shall obtain a negative result in the urine or serum pregnancy test performed within 3 days before the first dose of the investigational drug (cycle 1, day 1). If the urine pregnancy test result cannot be identified as negative, a blood pregnancy test is needed. Women of non-childbearing potential are defined as those who have not had menses for at least 1 year or who have undergone surgical sterilization or hysterectomy; 13. All subjects at risk of conception (including their partners) shall use contraceptives with an annual failure rate of less than 1% throughout the entire treatment period up to 120 days after the last dose of the investigational drug (or 180 days after the last dose of the chemotherapy drug).

Exclusion Criteria:

* 1. Diagnosed with malignant tumors other than non-small cell lung cancer within 5 years before the first dose, excluding radically cured cutaneous basal cell carcinoma, cutaneous squamous cell carcinoma, and/or radically resected carcinoma in situ; 2. Previously treated with selective FGFR inhibitors; 3. Have received any other investigational drug treatment or participated in another interventional clinical trial within 28 days before the first dose of the investigational drug, or have received anti-tumor drug treatment within 28 days before the first dose of the investigational drug (including Chinese herbal medicine with anti-tumor indications); 4. Have not recovered (i.e., reaching ≤ grade 1 or the baseline status, excluding asthenia and alopecia) from toxicity and/or complications caused by any intervention before the start of treatment; 5. With known symptomatic central nervous system metastasis and/or carcinomatous meningitis. Subjects with previously treated brain metastases are eligible if the disease is stable (no imaging evidence of progression in at least 4 weeks prior to the first dose of study treatment), there is no evidence of new or enlarging brain metastases on repeated imaging, and corticosteroids are not required in at least 14 days prior to the first dose of study treatment. Patients with carcinomatous meningitis should be excluded regardless of their clinically stability; 6. During pregnancy or lactation; 7. Known history of allotransplantation or allogeneic hematopoietic stem cell transplantation; 8. Subjects with abnormal laboratory parameters listed below:

  1. Serum phosphate > ULN;
  2. Serum calcium exceeds the normal range, or the calcium concentration corrected for serum albumin exceeds the normal range when serum albumin exceeds the normal range;
  3. Potassium level < lower limit of normal (LLN); potassium levels can be corrected by supplements at screening.

     9. With known history of human immunodeficiency virus (HIV) infection or confirmed with positive immune test results; 10. Presence of severe infection in the active phase or with poor clinical control; 11. Pleural effusion, ascites, or pericardial effusion with obvious clinical symptoms that require drainage; 12. Acute or chronic active hepatitis B or C infection; hepatitis B virus (HBV) DNA > 2000 IU/mL or 104 copies/mL; hepatitis C virus (HCV) RNA > 103 copies/mL; hepatitis B surface antigen (HbsAg) and anti-HCV antibody positive concurrently. Those who with relevant parameters lower than the above criteria after nucleotide antiviral treatment can be enrolled; 13. With clinically significant or uncontrolled heart diseases, including unstable angina, acute myocardial infarction within 6 months before the first dose, grade III/IV congestive heart failure (New York Heart Association), and uncontrolled arrhythmia (subjects with pacemakers or with atrial fibrillation but well controlled heart rate are allowed); 14. With ECG changes or medical history considered clinically significant by the investigator; QTcF interval > 480 ms at screening; for subjects with intraventricular conduction block (QRS interval > 120 ms), JTc interval can be used instead of QTc interval upon approval of the sponsor (in such cases, JTc must be ≤ 340 ms); 15. With uncontrolled hypertension (systolic pressure > 160 mmHg or diastolic pressure > 100 mmHg after the optimal medical treatment), or a history of hypertensive crisis or hypertensive encephalopathy; 16. With hepatic encephalopathy, hepatorenal syndrome, or liver cirrhosis with Child-Pugh grade B or C.

     17. Have received a major surgery (craniotomy, thoracotomy, or laparotomy) within 4 weeks prior to the first dose of study treatment, or will receive a major surgery during the study treatment period; 18. Pregnant or lactating women, or subjects expected to conceive or give birth during the study period from the screening visit to the completion of the safety follow-up visit (90 days after the last dose for male subjects); 19. Have received radiotherapy within 4 weeks before the first dose of the investigational drug. The subjects must be completely recovered from radiotherapy-related toxicity, with no need for corticosteroid treatment, and radiation pneumonitis must be excluded. For palliative radiotherapy for non-CNS diseases, a 2-week washout period is allowed; 20. Have a history of disorders of calcium and phosphorus metabolism or systemic electrolyte metabolism imbalance with ectopic calcification of soft tissues (excluding calcification of soft tissues such as skin, kidneys, tendon, or blood vessels without systemic electrolyte metabolism imbalance caused by injury, disease, and old age); 21. Clinically significant corneal or retinal diseases confirmed by ophthalmological examination; 22. Have used any potent CYP3A4 inhibitor (see Appendix A for details) or inducer within 14 days or 5 half lives (whichever is shorter) before the first dose of the investigational drug. Ketoconazole is allowed for external use; 23. With known allergic reactions to pemigatinib or excipients of pemigatinib; 24. Unable or unwilling to swallow pemigatinib or are suffering from significant digestive system diseases that may interfere with absorption, metabolism, or excretion; 25. Subjects with a history of vitamin D deficiency who require supraphysiological dose of vitamin D (except dietary vitamin D supplements); 26. Other acute or chronic diseases, psychiatric disorders, or laboratory abnormalities that may result in an increased risk associated with study participation or investigational drug administration or interfere with the interpretation of study results, and disqualify patients from the study in the investigator's judgment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-12-06 (Actual); Primary Completion 2023-12-06 (Estimated); Study Completion 2024-12-06 (Estimated)

PRIMARY OUTCOMES:
ORR | an expected average of 2 years
  ORR is defined as the proportion of subjects with complete response (CR) + those with partial response (PR) according to the RECIST1.1 criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, China

IPD SHARING:
Plan to Share IPD: Undecided